CLINICAL TRIAL: NCT06220773
Title: A Randomized, Double-blind, Multi-center, Phase 3 Study to Evaluate the Efficacy and Safety of BR1019A and BR1019B Combination Therapy in Patients With Essential Hypertension and Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Efficacy and Safety of BR1019A and BR1019B Combination Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FDC-CT-301
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Essential Hypertension; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Essential Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BR1019A + BR1019B + BR1019C-1 (Experimental)
  Interventions: Drug: BR1019A; Drug: BR1019B; Drug: BR1019C-1
- BR1019A + BR1019B-1 + BR1019C-1 (Active Comparator)
  Interventions: Drug: BR1019A; Drug: BR1019B-1; Drug: BR1019C-1
- BR1019A-1 + BR1019B + BR1019C-1 (Active Comparator)
  Interventions: Drug: BR1019B; Drug: BR1019A-1; Drug: BR1019C-1
- BR1019A-1 + BR1019B + BR1019C (Other)
  Interventions: Drug: BR1019B; Drug: BR1019C; Drug: BR1019A-1

INTERVENTIONS:
Drug: BR1019A — Subjects take the investigational products once a day for 12 weeks.
  Arms: BR1019A + BR1019B + BR1019C-1; BR1019A + BR1019B-1 + BR1019C-1
Drug: BR1019B — Subjects take the investigational products once a day for 12 weeks.
  Arms: BR1019A + BR1019B + BR1019C-1; BR1019A-1 + BR1019B + BR1019C; BR1019A-1 + BR1019B + BR1019C-1
Drug: BR1019C — Subjects take the investigational products once a day for 12 weeks.
  Arms: BR1019A-1 + BR1019B + BR1019C
Drug: BR1019A-1 — Subjects take the investigational products once a day for 12 weeks.
  Arms: BR1019A-1 + BR1019B + BR1019C; BR1019A-1 + BR1019B + BR1019C-1
Drug: BR1019B-1 — Subjects take the investigational products once a day for 12 weeks.
  Arms: BR1019A + BR1019B-1 + BR1019C-1
Drug: BR1019C-1 — Subjects take the investigational products once a day for 12 weeks.
  Arms: BR1019A + BR1019B + BR1019C-1; BR1019A + BR1019B-1 + BR1019C-1; BR1019A-1 + BR1019B + BR1019C-1

SUMMARY:
The objective of this clinical study is to Evaluate the Efficacy and Safety of BR1019A and BR1019B combination therapy in Patients with Essential Hypertension and Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Those with type 2 diabetes mellitus & essential hypertension
* Those who agree to discontinue existing antihypertensive and/or oral hypoglycemic drugs during the clinical trial
* Those who are judged medically reasonable by investigator to be able to discontinue existing antihypertensive and/or oral hypoglycemic drugs(except for Metformin) during the clinical trial

Exclusion Criteria:

* Those who meet the following criteria

  * Those with a history of secondary hypertension or suspected secondary hypertension; (Including but not limited to; e.g., renovascular disease, adrenal medullary and cortical hyperfunctions, coarctation of the aorta, primary hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromocytoma and polycystic kidney disease, etc.)
  * Those with clinical significant orthostatic hypotension accompanied by symptoms
  * Those with diabetes mellitus taking renin inhibitors(Aliskiren) or moderate to severe renal impairment
  * Those with diabetic nephropathy taking ACE inhibitors
  * Those with type 1 diabetes mellitus, secondary diabetes mellitus, severe insulin-dependent diabetes, diabetic ketoacidosis or lactic acidosis
  * Those with uncontrolled, severe diabetic complications (Micro-vascular complications(e.g., nephropathy, retinopathy, neuropathy, etc.), Macro-vascular complications)
  * Diabetic coma or pre-coma

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The change of mean sitting systolic blood pressure from baseline in BR1019A+BR1019B+BR1019C-1 at Week 12 compared to BR1019A-1+BR1019B+BR1019C-1 | 12 weeks from Baseline Visit
The change of HbA1c from baseline in BR1019A+BR1019B+BR1019C-1 at Week 12 compared to BR1019A+BR1019B-1+BR1019C-1 | 12 weeks from Baseline Visit

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No